CLINICAL TRIAL: NCT03892824
Title: Carotid Artery ImPlant for Trapping UpstReam Emboli (CAPTURE 2) for Preventing Stroke in Atrial Fibrillation Patients Taking Oral Anticoagulants
Brief Title: Carotid Artery Implant for Preventing Stroke in Atrial Fibrillation Patients Taking Oral Anticoagulants
Acronym: CAPTURE2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Javelin Medical (Industry)
Collaborators: Genae (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CL-326
Record Dates: First submitted 2019-03-21; First posted 2019-03-27 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: AF; Stroke; Filter; Emboli; Carotid; OAC
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vine™ Filter + OAC (Experimental): Vine™ Filter in each common carotid artery (CCA) with oral anticoagulant treatment (either vitamin K antagonist (VKA) or novel oral anticoagulant (NOAC)) for the duration of the study
  Interventions: Device: Vine™ Embolic Protection System

INTERVENTIONS:
Device: Vine™ Embolic Protection System — The system includes the implant and the Vine™ Inserter (inserter) manufactured by Javelin Medical LTD (Israel). The inserter comprises a Motor Unit and a Needle Unit ("Needle Unit") available in two sizes. The system is operable when the Needle Unit is loaded with the implant (labeled "Loaded Needle Unit") and connected to the Motor Unit. A flag indicating the needle orientation is attached to the needle luer. The implant is automatically deployed from the needle upon activation of the operating button.

SUMMARY:
This study will assess the safety and performance of the Vine™ Embolic Protection System (embolic filtering device) in atrial fibrillation (AF) patients on top of oral anticoagulants (OAC), and remain at high risk for stroke recurrence. All patients will receive bilateral implants in the common carotid arteries

DETAILED DESCRIPTION:
The Vine™ filter (Vine™ or implant) is a permanent carotid filter designed for stroke prevention in AF patients taking OAC at high stroke risk (CHA2DS2-VASc ≤ 4 and stroke history). This patient population accounts for ~20% of the entire AF population, which is ~300K/year in the United State and EU. The implant is designed to exclude emboli > 1.4mm in size from reaching the anterior circulation. In AF patients, approximately 80% of strokes are total or partial anterior circulation strokes caused by occlusions of the main branches of the Circle of Willis, mainly M1-2, and rarely A1-2. The diameter of these branches, in the majority of cases, is > 1.5 mm

ELIGIBILITY:
Inclusion Criteria:

* Documented AF
* CHA2DS2-VASc score ≥ 4 and history of ischemic stroke (including TIA with positive neuro-imaging)
* No contra-indication for patient to receive an OAC, either vitamin K antagonist (VKA) or novel oral anticoagulant (NOAC) for the duration of the study
* Age > 50 years
* Maximal (systolic) CCA diameter range: ≥ 4.8mm and ≤ 9.8mm
* CCA accessibility: up to 40mm from skin to CCA center, safe approach
* Implantation segment free of atherosclerotic disease as determined by ultrasound imaging
* Patient is able and willing to provide informed consent

Exclusion Criteria:

* Evidence of carotid stenosis > 30% [CCA, internal carotid artery (ICA), or external carotid artery (ECA)]
* Evidence of carotid dissection
* Pre-existing stent(s) in CCA
* Female who is pregnant or who is planning to become pregnant during the course of the study
* Life expectancy of less than two years
* Active systemic infection
* Known sensitivity to nickel or titanium metals, or their alloys
* Known hereditary or acquired coagulation disorders
* Any planned surgical or endovascular treatment within 30 days after the implantation procedure
* A co-morbid disease or condition that could confound the neurological and functional evaluations or compromise survival or ability to complete follow-up assessments* Current use or a recent history of illicit drug(s) use or alcohol abuse (defined as regular or daily consumption of more than four alcoholic drinks per day)
* Active participation in another investigational drug or device treatment study
* Inability to complete all scheduled follow-up
* Any other condition that in the opinion of the investigator may adversely affect the safety of the patient or would limit the patient's ability to complete the study
* History of intracerebral hemorrhage (ICH) and/or hemorrhagic stroke
* Event of stroke/TIA in the past 14 days

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2027-10-24 (Estimated)

PRIMARY OUTCOMES:
Number of participants that had Ischemic Stroke and/or Hemorrhagic stroke and/or implantation procedure complications | 30 days from implantation procedure
  Major Adverse Events (MAEs) within 30 days of the final index (implantation) procedure, defined as the composite that includes any of the following:
  * Any ischemic stroke with ischemic foci confined to the territories of Vine™ implanted arteries
  * Hemorrhagic stroke or major hemorrhage while receiving additional antithrombotic therapy required for Vine™ implantation
  * Any Vine™ or Vine™ implantation procedure-related complication that requires surgery or endovascular treatment, or results in death or major disability

SECONDARY OUTCOMES:
Number of participants that had Ischemic Stroke and/or Hemorrhagic stroke and/or Device complications. | one and two years from implantation procedure
  * Any ischemic stroke with ischemic foci confined to the territories of Vine™ implanted arteries
  * Hemorrhagic stroke or major hemorrhage while receiving additional antithrombotic therapy required for Vine™ implantation
  * Any Vine™ or Vine™ implantation procedure-related complication that requires surgery or endovascular treatment, or results in death or major disability
Number of properly positioned implants | 30 days from implantation procedure
  proper implant position in each common carotid artery (CCA)
Number of participants that had disabling strokes | 30 days, one and two years from implantation procedure
  Disabling stroke
Number of Implantation success | immediately after the procedure
  implantation attempt resulting in proper implant position immediately after the procedure without any device/procedure related complication that requires surgery or endovascular treatment for correction, or that results in death or major disability
Number of properly positioned implants | one and two years from implantation procedure
  Proper implant position in each CCA
Number of observed thrombi on the device | 30 days, one and two years from implantation procedure
  Thrombus on implant detected by ultrasound imaging
Number of death cases | one and two years from implantation procedure
  Death
Number of strokes (any kind) | one and two years from implantation procedure
  Total number of strokes

CONTACTS AND LOCATIONS:
Locations (17):
- Belgium (2):
  - OLV Ziekenhuis, Aalst
  - ZNA Stuivenberg, Antwerp
- Na Homolce Hospital, Prague, Czechia
- Germany (3):
  - Alfried-Krupp Krankenhaus Rüttenscheid, Essen
  - Cardio Vasculäres Centrum Frankfurt, Frankfurt
  - Cardioangiologisches Centrum Bethanien, Frankfurt
- Greece (4):
  - General Hospital of Athens "Hippokrateio", Athens
  - Laiko Hospital, Athens
  - University General Hospital of Larisa, Larissa
  - European Interbalkan Medical Center, Thessaloniki
- Gottsegen György Hungarian Institute of Cardiology, Budapest, Hungary
- Israel (4):
  - Carmel, Haifa
  - Shaari Tzedek, Jerusalem
  - Rabin Medical Center (RMC), Petah Tikva
  - Poria, Tiberias
- Szpital Kliniczny Przemienienia Pańskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Pracownia Hemodynamiki Serca, Poznan, Poland
- Hospital Universitario Ramon y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No